CLINICAL TRIAL: NCT01550952
Title: Interscalene Dynamometer Pilot Study
Status: Completed | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-002
Record Dates: First submitted 2012-03-01; First posted 2012-03-12 (Estimated); Results first posted 2016-03-31 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2012-09

CONDITIONS: Total Shoulder Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Total shoulder arthroplasty (shoulder replacement) can cause severe postoperative pain. Commonly, patients receive general anesthesia with interscalene block (injection of local anesthetic or numbing medicine near nerves in the shoulder) during surgery. As a result of the interscalene block, patients often experience sensory and motor blockade. The purpose of this study is to determine the effects of the interscalene block on the anterior deltoid muscle and hand grip strength after total shoulder arthroplasty.

DETAILED DESCRIPTION:
Total shoulder arthroplasty can cause severe postoperative pain. Pain management includes general anesthesia with interscalene block during surgery and intravenous (IV) hydromorphone patient controlled analgesia (PCA) and oral opioid analgesics given after surgery. Side effects, such as motor blockade, may impair participation in physical therapy and diminish patient satisfaction. In order to prepare for a future study that will examine what mixtures of adjuncts/additives will best prevent recovery room pain and minimize motor blockade, the investigators are conducting this pilot study to collect preliminary data on current practice. The investigators believe the current regimen will provide adequate pain relief, but may cause extensive motor blockade and reduce patients' muscle strength after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for primary total shoulder arthroplasty
* Age 18 to 80 years old
* Planned use of general anesthesia via laryngeal mask airway (LMA) and peripheral nerve block
* Ability to follow study protocol
* Patients with American Society of Anesthesiologists (ASA) physical status of I, II or III

Exclusion Criteria:

* Patients younger than 18 years old and older than 80
* Patients not intending to receive general anesthesia and peripheral nerve block
* Allergy or intolerance to one of the study medications
* Patients with an ASA of IV
* Hepatic or renal insufficiency
* Chronic opioid use (taking opioids for longer than 3 months)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18-80 years old who are undergoing primary total shoulder arthroplasty.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques T YaDeau, MD, PhD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Total Shoulder Arthroplasty Patients
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Total Shoulder Arthroplasty Patients
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 10
Body Mass Index [Number; unit: participants]
  Normal | 1
  Overweight | 3
  Obese | 6

OUTCOME MEASURES:

1. Primary Outcome: Anterior Deltoid Strength
Description: Anterior deltoid strength as measured by a dynamometer. Percentage change in measure as compared to post-surgery (with post-surgery measure at 0%).
Time Frame: 2 days postoperatively
Population: One participant declined assessment due to soreness in the shoulder muscle.
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Total Shoulder Arthroplasty Patients
Number analyzed (Participants) | 9
percent | 77 [52 to 119]

2. Primary Outcome: Hand Grip Strength
Description: Hand grip strength as measured by a dynamometer. Percentage change in measure as compared to post-surgery (with post-surgery measure at 0%).
Time Frame: 2 days postoperatively
Population: One participant declined assessment due to soreness in the shoulder muscle.
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Total Shoulder Arthroplasty Patients
Number analyzed (Participants) | 9
percent | 90 [76 to 99]

3. Secondary Outcome: Number of Participants With Reduced Sensation in a Dermatome
Description: Pin-prick sensation assessed.
Time Frame: 2 days postoperatively
Population: Dermatomes could not be assessed for one patient due to sedation
Measure: Number; unit: participants
Arm/Group | Total Shoulder Arthroplasty Patients
Number analyzed (Participants) | 9
participants | 8

4. Secondary Outcome: Numeric Rating Scale (NRS) Pain Scores With Movement
Description: NRS pain scores (0-10; 0 = no pain, 10 = worst pain possible) assessed.
Time Frame: 2 days postoperatively
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Total Shoulder Arthroplasty Patients
Number analyzed (Participants) | 10
units on a scale | 0.8 [0 to 1.5]

5. Secondary Outcome: Total Oral Opioid Intake in 48hrs
Description: Opioid Usage
Time Frame: 0-48hrs
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Total Shoulder Arthroplasty Patients
Number analyzed (Participants) | 10
mg | 52.3 (32.7)

ADVERSE EVENTS:
Arm/Group | Total Shoulder Arthroplasty Patients
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes